CLINICAL TRIAL: NCT03185767
Title: Long Non Coding RNA IN Systemic Lupus
Brief Title: Long Non Coding RNA in Complications of Systemic Lupus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mai ahmec, teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 12345SLE
Record Dates: First submitted 2017-06-03; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Complication in Systemic Lupus Erythematosus
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLE group (Other)
  Interventions: Other: blood sampling
- control group (Other)
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — blood sampling

SUMMARY:
the precise role of RNA in setting of this complication in systemic lupus erythematosus (SLE) is largely unknown

ELIGIBILITY:
Inclusion Criteria:

* with systemic lupus

Exclusion Criteria:

vasculitis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-07-01 (Estimated)

PRIMARY OUTCOMES:
non coding RNA expression by real time PCR | 1 year
  non coding RNA expression by real time PCR to evaluate thier role in lupus

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No